CLINICAL TRIAL: NCT03173222
Title: A Clinical Study of Electroacupuncture for Abdominal Pain Relief in Patients With Acute Pancreatitis
Brief Title: Electroacupuncture for Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DongGuk University (Other)
Responsible Party: Principal Investigator, Dong Kee Jang, Assistant professor, DongGuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HI16C0887
Record Dates: First submitted 2017-05-30; First posted 2017-06-01 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- EA1 (Active Comparator)
  Interventions: Procedure: Electroacupuncture
- EA2 (Active Comparator)
  Interventions: Procedure: Electroacupuncture
- Control (No Intervention)

INTERVENTIONS:
Procedure: Electroacupuncture — A combined procedure with acupuncture and electric current stimulation. Local electroacupuncture will be given in group EA 1, while local with distal electroacupuncture will be given in group EA 2.
  Arms: EA1; EA2

SUMMARY:
This study aims to prove the efficacy of electroacupuncture (EA) for pain relief in patients with acute pancreatitis compared with conventional treatment. Patients diagnosed with acute pancreatitis will be enrolled after obtaining informed consents. They will be randomly assigned to EA 1, EA 2, or control group in a 1:1:1 ratio. All the enrolled patients will basically receive the conventional standard-of-care therapy for acute pancreatitis. Local electroacupuncture will be given in group EA 1, while local with distal electroacupuncture will be given in group EA 2, additionally. For the conventional therapy, first non-steroidal anti-inflammatory drugs will be administered; afterwards, if inadequately controlled, low-potency narcotic analgesics such as codeine and then high-potency narcotic analgesics such as morphine or meperidine will be given sequentially as required. The patients randomized to the EA 1 and 2 groups will undergo 1 session of electroacupuncture daily from day 1 until day 4, or until pain is resolved. The primary endpoint is the visual analogue scale (VAS) for pain on day 5. Secondary endpoints include daily VAS, requirement of analgesics, changes of inflammatory markers, and hospital days.

DETAILED DESCRIPTION:
Acute pancreatitis (AP) causes significant abdominal pain, which can destroy patients'quality of life. Most patients have associated nausea and vomiting. Pain control for such patients is the mainstay of AP management. Opioids are safe and effective for pain control in patients with AP. Compared with other analgesic options, opioids may decrease the need for supplementary analgesia. However, frequent administration of opioid analgesics may result in opioid dependency. Unfortunately, any innovative treatment for the pain better than opioids has not been developed in the medical science so far. Therefore, the development of novel treatment for pain relief without triggering dependency is urgent. Acupuncture originated in China approximately 2000 years ago and is one of the oldest medical procedures in the world. Acupuncture continued to be developed and codified in texts over the subsequent centuries and gradually became one of the standard therapies used in China. Later, acupuncture was introduced to other countries including Asia, Europe, and Unites States. The most thoroughly studied application of acupuncture is for pain relief. In this sense, acupuncture in the oriental medicine could be an appropriate alternative for opioid analgesics, since it has been known as an effective treatment for pain relief without dependency. Electroacupuncture (EA) is a form of acupuncture where a small electric current is passed between pairs of acupuncture needles. Previous studies suggested that EA blocks pain by activating a variety of bioactive chemicals through peripheral, spinal, and supraspinal mechanisms. Therefore, we plan to prove the efficacy of EA for pain relief in patients with AP compared with conventional treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute pancreatitis
* The definition of acute pancreatitis is based on the fulfillment of 2 out of 3 of the following criteria: clinical (upper abdominal pain), laboratory (serum amylase or lipase > 3 x upper limit of normal) and/or imaging (computed tomography, magnetic resonance imaging, ultrasonography) criteria.

Exclusion Criteria:

* Those whose informed consent could not be obtained
* Patients with severe pancreatitis accompanying multiple organ failure

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-08-29 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale of pain | Day 5 (after planned interventions)
  0-100

CONTACTS AND LOCATIONS:
Locations (1):
- Dongguk University Ilsan Medical Center, Goyang-si, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ng SSM, Leung WW, Mak TWC, Hon SSF, Li JCM, Wong CYN, Tsoi KKF, Lee JFY. Electroacupuncture reduces duration of postoperative ileus after laparoscopic surgery for colorectal cancer. Gastroenterology. 2013 Feb;144(2):307-313.e1. doi: 10.1053/j.gastro.2012.10.050. Epub 2012 Nov 6. PMID 23142625
- [Derived] Kee Jang D, Kyu Lee J, Yung Jung C, Ho Kim K, Ra Kang H, Sun Lee Y, Hwa Yoon J, Ro Joo K, Kyu Chae M, Hyeon Baek Y, Seo BK, Hyub Lee S, Lim C. Electroacupuncture for abdominal pain relief in patients with acute pancreatitis: A three-arm randomized controlled trial. J Integr Med. 2023 Nov;21(6):537-542. doi: 10.1016/j.joim.2023.10.004. Epub 2023 Nov 2. PMID 37973472
- [Derived] Jang DK, Jung CY, Kim KH, Lee JK. Electroacupuncture for abdominal pain relief in patients with acute pancreatitis: study protocol for a randomized controlled trial. Trials. 2018 May 16;19(1):279. doi: 10.1186/s13063-018-2644-1. PMID 29769133